CLINICAL TRIAL: NCT07157150
Title: The Effects of Rule Modifications in 3v3 and 4v4 Small-Sided Games on Cardiovascular and Technical Performance in Elite Football Players
Acronym: CARDIO-TECH SS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamza Kucuk (Other)
Responsible Party: Sponsor-Investigator, Hamza Kucuk, Assoc Prof., Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HKucuk-SSG-2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Exercise Training; Exercise Physiology
Keywords: Small sided games; physiological responses; lactate concentration; heart rate dynamics; aerobic capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Play (Experimental): Elite football players participate in 3v3 and 4v4 small-sided games without restrictions, allowing free play conditions.
  Interventions: Behavioral: Free Play SSG
- Controlled Pass (Experimental): Elite football players participate in 3v3 and 4v4 small-sided games where a minimum number of passes is required before attempting to score.
  Interventions: Behavioral: Controlled Pass

INTERVENTIONS:
Behavioral: Free Play SSG — Other current and former name(s) or alias(es), if any, different from the Intervention Name(s), that the sponsor has used publicly to identify the intervention(s), including, but not limited to, past or present names such as brand name(s), or serial numbers
  Arms: Free Play
Behavioral: Controlled Pass — Participants train in 3v3 and 4v4 football games under Controlled Pass rules for 8 weeks.
  Arms: Controlled Pass

SUMMARY:
This study explores how different small-sided football games affect players' heart and technical skills. We will compare two ways of playing: "Free Play," where players act freely, and "Controlled Pass," where passing rules are used. Elite football players will participate in both types of games on small fields (3 vs 3 and 4 vs 4). We will measure heart responses (like heart rate) and how often players touch the ball. The goal is to help coaches choose the best game format to improve fitness and technical ability in training.

DETAILED DESCRIPTION:
Small-sided games (SSGs) are widely used in football training because they combine technical, tactical, and physical demands in a single activity. However, the way rules are modified during these games can change how players respond both physiologically and technically. Despite the popularity of SSGs in elite football, limited evidence exists regarding how specific rule modifications influence cardiovascular strain and technical involvement in real training settings.

This study was designed to examine the effects of two rule conditions, Free Play and Controlled Pass, in both 3v3 and 4v4 SSG formats. The Free Play condition allows players to participate without additional restrictions, whereas the Controlled Pass condition requires a minimum number of passes before attempting to score. These modifications are expected to alter both the cardiovascular responses and technical actions of players.

A total of 24 elite male football players, aged 18 to 30 years, with at least five years of professional experience, were recruited to participate. All participants underwent baseline assessments and were then assigned to play both conditions in a randomized sequence. Each SSG session lasted eight weeks and was closely monitored by the research team. Heart rate responses were measured continuously using Polar heart rate monitors, and technical performance was evaluated through video-based notational analysis.

The primary outcomes of interest were maximum heart rate (HRmax) and percentage of HRmax, which provide indicators of cardiovascular load. The secondary outcomes were the number of ball touches, reflecting the degree of technical involvement during play. Statistical analysis included paired-samples t-tests and Wilcoxon signed-rank tests, with significance set at p < 0.05.

Preliminary evidence suggests that Free Play conditions elicit greater cardiovascular load, especially in the initial sets of training, while Controlled Pass conditions promote higher technical engagement by increasing ball touches. The findings are expected to help coaches and practitioners make evidence-based decisions when designing training tasks for elite football players. Specifically, coaches may select Free Play conditions when the aim is to maximize physical conditioning and Controlled Pass rules when the aim is to enhance technical and tactical involvement.

This study was approved by the Ethics Committee of Bilecik Şeyh Edebali University (approval date: June 29, 2020; decision no: 8/26). All participants provided written informed consent prior to enrollment, and the study was conducted in accordance with the Declaration of Helsinki.

By addressing the gap in evidence on rule modifications in SSGs, this trial provides new insights into optimizing training design for elite football. Its findings may inform practical applications for strength and conditioning coaches, sport scientists, and football practitioners worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Male elite football players
* Aged 18-30 years
* At least 5 years of professional football experience
* Currently training and competing at the professional level

Exclusion Criteria:

* Presence of cardiovascular, respiratory, or musculoskeletal disease or injury that could interfere with participation
* Use of medication affecting cardiovascular function
* Inability to complete training sessions or follow study protocol
* Refusal to provide informed consent

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum Heart Rate (HRmax) | During 8 weeks of training sessions
  HRmax recorded continuously using Polar heart rate monitors during 3v3 and 4v4 small-sided games under Free Play and Controlled Pass conditions.
Percentage of Maximum Heart Rate (%HRmax) | During 8 weeks of training sessions
  Relative cardiovascular load calculated as percentage of HRmax, measured via Polar HR monitors across Free Play and Controlled Pass sessions.

SECONDARY OUTCOMES:
Number of Ball Touches | During 8 weeks of training sessions
  Technical performance indicator measured by video-based notational analysis of each participant's ball contacts during 3v3 and 4v4 games.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (e.g., age, heart rate responses, ball touches) that underlie the results of the study will be shared. Supporting documents, including the study protocol and statistical analysis plan, will also be available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the main results and ending 3 years after publication.
Access Criteria: Researchers who provide a methodologically sound proposal for use in achieving the aims of their research will be granted access. Proposals should be directed to [your institutional email]. Data will be shared via secure data repository.

REFERENCES:
- [Background] Şar, H., Çelgin, G. S., Arslanoğlu, C., Kızılörs, G., Arslanoğlu, E., Ceylan, L., & Küçük, H. (2025). The Effects of FIFA 11+ and Harmoknee Warm-Up Protocols on Flexibility, Vertical Jump and Shooting Speed in Female Football Players: A Comparative Study. Applied Sciences, 15(9), 4936. https://doi.org/10.3390/app15094936